CLINICAL TRIAL: NCT05497908
Title: Transverse Abdominis Plane (TAP) Block in EXtreme Lateral Interbody Fusion (XLIF) Surgery: a Pilot Feasibility Trial
Brief Title: Feasibility of TAP for XLIF Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Stafmember Anesthesiology and Intensive Care, Head of Science department Anesthesiology and Intensive Care, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: f/2022/050
Record Dates: First submitted 2022-07-28; First posted 2022-08-11 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Pain, Postoperative
Keywords: eXtreme Lateral Interbody Fusion (XLIF) surgery; transversus abdominis plane (TAP) block
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transversus abdominis plane (TAP) block via lateral approach (Experimental): This group receives a Transversus abdominis plane (TAP) block via lateral approach
  Interventions: Procedure: TAP block via lateral approach
- Transversus abdominis plane (TAP) block via posterior approach (Experimental): This group receives a Transversus abdominis plane (TAP) block via posterior approach
  Interventions: Procedure: TAP block via posterior approach
- Control group (No Intervention): The control group receives no TAP block.

INTERVENTIONS:
Procedure: TAP block via lateral approach — TAP block via lateral approach
  Arms: Transversus abdominis plane (TAP) block via lateral approach
Procedure: TAP block via posterior approach — TAP block via posterior approach
  Arms: Transversus abdominis plane (TAP) block via posterior approach

SUMMARY:
Key questions of this feasibility trial will be the feasibility of performing the TAP block in XLIF patients, screen for safety of the block and preliminary investigate the influence on pain control and quality of recovery. The investigators hypothesize that visualization of lateral TAP will be superior to visualization of posterior TAP, protocol adherence and safety profile to be excellent and both blocks to be superior in terms of analgesia compared to no block.

DETAILED DESCRIPTION:
Enhanced recovery after surgery trajectories have been widely adopted after its first publications mentioned faster recovery and better patient outcomes whilst reducing costs . The recent COVID pandemic further emphasized the importance of reducing hospital length of stay for elective procedures, both from a patient quality as from an economic point of view. Minimally invasive surgical techniques are key in allowing enhanced recovery after surgery programs: eXtreme Lateral Interbody Fusion (XLIF) is one of those surgical techniques. XLIF has a reported enhanced recovery with a short hospital stay. On the other hand, multimodal anesthetic regimens with the potential to reduce the need for long-acting opioids are crucial in supporting early recovery after surgery. Regional anesthesia is an important element in multimodal analgesia. It has a significant effect on acute pain and reduces morphine consumption. Opioid sparing regional techniques obviously reduce opioid side effects leading to less postoperative nausea and vomiting (PONV), pruritus and drowsiness. Despite the increasing evidence for locoregional anesthetic techniques in enhanced recovery after surgery trajectories, the quest for the ideal regional technique, timing of block placement, local anesthetic and single shot versus catheter often remains a challenge. Traditional locoregional anesthetic techniques and spine surgery have known a reluctant relationship. Spine surgeons typically prefer optimal conditions for a decent neurologic examination after the surgical procedure to recognize early surgical complications. Classic neuraxial analgesia and peripheral nerve blocks might compromise this clinical neurologic follow-up. On the other hand, anesthetic guidelines raise concerns about the safety of locoregional anesthesia in patients with existing neurologic disease as neurologic conditions might worsen, especially after suboptimal application of locoregional techniques. However, during the last decade the practice of locoregional anesthesia expanded with the introduction of multiple planar blocks. In these blocks, local anesthetics are injected in a plane -usually an intermuscular plane- providing anesthesia to performant sensory nerve branches without affecting the motor function of the nerves. Clinically, in uttermost plane blocks a sensory blockade is achieved without the loss of ambulation. The thoracolumbar interfascial plane (TLIP) block and erector spinae block (ESB) were the first plane blocks to be introduced in spine surgery. A systematic review on the use of TLIP in back surgery found a significant lower use of perioperative opioids and PONV compared to no block or wound infiltration, as well as significantly lower postoperative pain scores compared to no block. However, concerns on blinding and a high allocation bias compromise the generalizability of this systematic review. The TLIP block also includes the risk for neuraxial injury and is a technically challenging block placed with the patient in uncomfortable prone position. Furthermore, the site of injection interferes with the corresponding surgical field. Therefore, some centers started performing the ESB for spine surgery. In a multicenter, non-blinded prospective trial a significant reduction in pain but not in opioid-consumption after bilateral ESB for major decompressive spine surgery was found. A retrospective case-matched study also found a reduction in pain scores and hospital length of stay but not in opioid use after posterior lumbar interbody fusion (PLIF). A blinded RCT in the Chinese population did find a significant reduction in pain scores and opioid requirements after lumbar fusion surgery. However, in this study the ESB was placed at a lower than conventional lumbar two (L2) level. This is important since the local anesthetics injected in the erector spinae plane spread towards the paravertebral and epidural spaces, targeting both the dorsal and ventral rami of the spinal nerve. Albeit, the ESB may affect motor function of the nerves in the surgical area, potentially interfering with intraoperative neuromonitoring as well as postoperative clinical neurologic examination. During XLIF surgery, indeed neuromonitoring is required to ensure a safe working corridor in relation to the lumbosacral plexus. Sofin et al. introduced the transversus abdominis plane (TAP) block for lumbar spine fusion via a lateral (LLIF) and anterior (ALIF) approach. In a feasibility trial, all patients received the block and no block-related adverse events were noted. The TAP block has been shown to be effective when used as an adjunct in multimodal analgesic strategies after abdominal surgery. First described by Rafi in 2001, the TAP block evolved from a blind landmark technique to an ultrasound-guided technique with subcostal and posterior variations. The abdominal wall block is achieved by injecting a high-volume, low concentration mixture of local anesthetics selectively between the interior and exterior abdominal muscles. Cadaver studies in which dye was injected found spread of the dye between the iliac crest, costal margin and rectus muscle with an average area of 45cm2. Additional MRI studies found retrograde spread of contrast to the paravertebral spaces between T4 and L1 when the TAP landmark technique and ultrasound-guided posterior approach were used. This in contrast to the subcostal and lateral TAP block where the spread pattern was confined to the anterior abdominal wall. Clinically, TAP block has been proven to be superior to placebo after a variety of abdominal surgeries such as inguinal hernia repair, open appendectomy, laparoscopic cystectomy and cesarean section. Furthermore, TAP catheters have shown non-inferiority for pain scores compared to epidural catheters after open renal and hepatobiliary surgery . Importantly, in these abdominal surgeries most patients still required some opioids for visceral analgesia. Therefore, experts suggest short stay procedures with the least visceral manipulation benefit most from single show abdominal wall blocks. The XLIF procedure might be an excellent indication for this TAP block since peritoneal manipulation is avoided in this surgical procedure. Last year, the earlier cited group by Sofin performed a retrospective study in 250 patients to investigate associations between TAP block and outcomes after LLIF/ALIF. They found a significantly shorter hospital length of stay (LOS) with TAP block after multivariate analysis. Opioid consumption and pain scores did not differ significantly. However, in the TAP group, a significantly larger proportion of patients had ALIF surgery. By consequence, the authors might not just have compared block versus no block but also have compared two types of surgery.

The effectiveness of TAP blocks on ALIF surgery is not unsurprising since the incision of ALIF surgery is fully comparable to the incision made during a cesarean section or to a surgical access for the lower abdominal region. To investigate the influence on outcome of TAP block after XLIF surgery however, the investigators will perform a prospective, randomized feasibility trial. Patients will be randomized on a 1:1:1 ratio in to three groups: lateral TAP block, posterior TAP block and no block. Key questions of this feasibility trial will be the feasibility of performing the TAP block in XLIF patients, screen for safety of the block and preliminary investigate the influence on pain control and quality of recovery. The investigators hypothesize visualization of lateral TAP will be superior to visualization of posterior TAP, protocol adherence and safety profile to be excellent and both blocks to be superior in terms of analgesia compared to no block.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

  * Scheduled for elective lumbar XLIF surgery

    * 1 level
    * multilevel
  * Patient being able to give informed consent
  * Patient being able to understand and use the PCIA system
  * Body Mass Index (BMI) ≤ 35 kg/m2

Exclusion Criteria:

* - Refusal to participate
* Chronic strong opioid use (WHO analgesic ladder step 3)
* Allergy to local anesthetics
* Antecedents of lumbar back surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Identification rate of the correct transverse abdominis plane block | immediately after the surgery
  Identification rate of the correct transverse abdominis plane block by ultrasound as assessed by a five-point-scale which can be found as supplement (very good -good - acceptable -poor - very poor)

SECONDARY OUTCOMES:
Total morphine consumption | 12 hours after surgery
  Total morphine consumption by PCIA < 12 hours after the end of surgery
Patient recruitment rate | through study completion, an average of 1 year
  ratio of patients giving informed consent to the number of eligible patients who were approached to participate
Adherence rate to protocol | 12 hours after surgery
  number of patients who completed correct follow-up until 12h after surgery
total operation room time | during the surgery
  evaluation of the total operation room time
Assessment of the number of patients with local anesthestia systemic toxicity (LAST) | during the stay at the PACU
  Assessment of the number of patients with local anesthestia systemic toxicity (LAST) at the postoperative care unit (PACU): perioral numbness, metallic taste, tinnitus, convulsion, bradycardia < 40 beats per minute. This evaluation will be performed by a physician who will examine the patients for these symptoms
Number of patients in need of additional analgesic drugs at PACU | during the stay at the PACU
  Number of patients in need of additional analgesic drugs at PACU such as morphine or clonidine
Incision region pain scores | at baseline and at 4, 8, 12 and 24 hours after surgery
  evaluation of the Incision region pain scores with an 11 point numerical scale (NRS) with 0 indicating no pain and 10 indicating worst imaginable pain
Lumbar back pain scores | at baseline and at 4, 8, 12 and 24 hours after surgery
  evaluation of the lumbar back pain scores with an 11 point numerical scale (NRS) with 0 indicating no pain and 10 indicating worst imaginable pain
time to first mobilisation | immediately after the surgery until postoperative day 3
  evaluation of time to first mobilisation
quality of recovery | postoperative day 3
  evaluation of the Quality of recovery measured by the Quality-of-Recovery-40 (QoR 40) scale on postoperative day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No